CLINICAL TRIAL: NCT03048877
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Apatinib in Locally Advanced or Metastatic Radioactive Iodine-refractory Differentiated Thyroid Cancer
Brief Title: Efficacy of Apatinib in Radioactive Iodine-refractory Differentiated Thyroid Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Yansong Lin, Prof. M.D., Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PUMCH-NPLA81H-Ahead-T302
Record Dates: First submitted 2017-02-03; First posted 2017-02-09 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Differentiated Thyroid Cancer
Keywords: Radioactive iodine-refractory; differentiated thyroid cancer; Apatinib; anti-angiogenesis drugs
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib (Experimental): Apatinib Mesylate Tablets
  Interventions: Drug: Apatinib Oral Tablet
- Placebo (Placebo Comparator): Placebo Tablets
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Apatinib Oral Tablet — Apatinib Mesylate Tablets
  Arms: Apatinib
Drug: Placebo Oral Tablet — Placebo Oral Tablet
  Arms: Placebo

SUMMARY:
Radioactive iodine-refractory differentiated thyroid cancer (RAIR-DTC) is a great challenge in the treatment of thyroid cancer. Tyrosine kinase inhibitors (TKIs), like sorafenib and lenvatinib which have been approved by food and drug administration (FDA), could not be affordable for most of the Chinese patients. Apatinib is a highly selective VEGFR2 inhibitor and reduces the angiogenesis of tumor effectively, which is a proven and effective drug in many solid tumors. A phase II study aims to assess the efficacy and safety of apatinib in RAIR-DTC ,which enrolled 20 patients and 10 of them had obtained a shout-term efficacy, demonstrating the peculiar potential in treatment of RAIR-DTC. In this study, the investigators aim to further explore the efficacy and safety of apatinib in RAIR-DTC.

DETAILED DESCRIPTION:
Primary Outcome Measure: Progression free survival of apatinib in RAIR-DTC.

Secondary Outcome Measures: Disease control rate, objective response rate, duration of response, changes of Tg and TgAb level in serum, overall survival, side effects and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Aged after 18 years (18 is included).
2. Locally advanced or metastatic differentiated thyroid cancer (papillary, follicular, Hurthle cells, poorly differentiated carcinoma). At least one measurable lesion (helical CT scan long diameter ≥10mm, meet the requirements of the standard Response Evaluation Criteria In Solid Tumors（RESCIST） version 1.1).
3. Disease progression within 12 months before inclusion.
4. Subjects must be 131I-refractory / resistant as defined by at least one of the following;

   * Lesions that do not demonstrate iodine uptake on any radioiodine scan;
   * Subjects received a single radioactive iodine therapy within 12 months (≥ 3.7 Giga Bequerel（GBq）[≥ 100 millicurie（mCi）]) and target lesion disease progression;
   * Every two radioactive iodine treatment interval <12 months, doses ≥ 3.7 GBq [≥100mCi], disease progress more than 12 months after at least once iodine therapy;
   * Received a total dose of radioactive iodine therapy ≥ 22.2 GBq (≥ 600 mCi);
5. Normal main organ function:

   * HB ≥ 90g / L;
   * ANC ≥1.5×109/L;
   * PLT ≥80×109/L;
   * BIL <1.5 × ULN;
   * ALT and AST <2.5 × ULN;
   * Cr≤1×ULN;
6. Eastern Cooperative Oncology Group（ECOG）Performance Status（PS） :0-2.
7. An expected survival of ≥ 3 months.
8. Pregnancy test (serum) has to be performed for woman of childbearing age within 7 days before enrolment and the test result must be negative. They shall take appropriate methods for contraception during the study until the 8th week post the last administration of study drug. For men, (previous surgical sterilization accepted), shall agree to take appropriate methods of contraception during the study until the 8th week post the last administration of study drug.
9. Patient has to voluntarily join the study and sign the Informed Consent Form for the study.
10. Good compliance is expected, according to the program requirements follow-up and recorded adverse reactions.

Exclusion Criteria:

1. Other thyroid cancer histological subtypes (such as medullary carcinoma, lymphoma or sarcoma).
2. Received VEGFR inhibitor (such as vandetanib, cabozantinib, lenvatinib, sunitinib, sorafenib, etc.) treatment within 1 months.
3. Subjects with poor-controlled arterial hypertension (systolic blood pressure> 140 mmHg and diastolic blood pressure > 90 mm Hg) despite standard medical management; coronary heart disease greater than Class II; II-level arrhythmia (including QT interval prolongation, for man ≥ 450 ms, for woman ≥ 470 ms) together with Class II cardiac dysfunction.
4. Factors that could have an effect on oral medication (such as inability to swallow, nausea, vomiting, chronic diarrhea and intestinal obstruction).
5. Subjects with high gastrointestinal bleeding risk, including the following conditions: local active ulcer lesions with positive fecal occult blood test (++); history of black stool, or vomiting blood in the past 3 months.
6. Abnormal Coagulation (INR>1.5、APTT>1.5 UNL), with tendency of bleed.
7. Disposition evidence of thrombosis/bleeding in 2 month (despite severity), hemoptysis in 2 months (bright red blood, 1/2 teaspoon).
8. Arterial /venous thromboembolic events, such as cerebrovascular accident, deep vein thrombosis and pulmonary embolism in the past 12 months.
9. Factors that could received radiotherapy or major surgery for anti - thyroid cancer in the past 28 days.
10. Factors that could received surgery (allows the full-recovery wound) or active hemorrhage, ulceration, intestinal perforation or intestinal obstruction in the past 28 days.
11. Uncontrolled infection.
12. Pregnant or lactating women.
13. Disposition evidence of depressive disorder (HAMD score ≥17).
14. Other conditions regimented at investigators' discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 24 months
  Progression free survival

SECONDARY OUTCOMES:
DCR | 24 months
  Disease control rate
ORR | 24 months
  Objective response rate
DoR | 24 months
  Duration of response
Changing trend of Tg and TgAb level in serum | 24 months
  Monitor the changes of Tg and TgAb level in serum regularly ( every 2~8 weeks, and addition examinations were needed if the participants' condition changed ) and draw the relevant changing curve to monitor the change of disease.
OS | 24 months
  Overall survival
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 24 months
  Record the number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Nanjing PLA 81 Hospital, Nanjing, Jiangsu
  - Peking Union Medical College Hospital, Beijing

REFERENCES:
- [Derived] Sun D, Zhang X, Jin X, Shi C, Sun Y, Zhang Y, Liang J, Lin Y. BRAFV600E mutation is associated with better prognoses in radioactive iodine refractory thyroid cancer patients treated with multi-kinase inhibitors: a retrospective analysis of registered clinical trials. Thyroid Res. 2025 Feb 10;18(1):5. doi: 10.1186/s13044-025-00223-0. PMID 39924483
- [Derived] Zhu Y, Liu K, Wang K, Peng L. Vascular Endothelial Growth Factor Receptor Inhibitors in Chinese Patients With Advanced Radioactive Iodine-Refractory Differentiated Thyroid Cancer: A Network Meta-Analysis and Cost-Effectiveness Analysis. Front Endocrinol (Lausanne). 2022 Jul 14;13:909333. doi: 10.3389/fendo.2022.909333. eCollection 2022. PMID 35909569
- [Derived] Lin Y, Qin S, Li Z, Yang H, Fu W, Li S, Chen W, Gao Z, Miao W, Xu H, Zhang Q, Zhao X, Bao J, Li L, Ren Y, Lin C, Jing S, Ma Q, Liang J, Chen G, Zhang H, Zhang Y, Zhou X, Sang Y, Hou Z. Apatinib vs Placebo in Patients With Locally Advanced or Metastatic, Radioactive Iodine-Refractory Differentiated Thyroid Cancer: The REALITY Randomized Clinical Trial. JAMA Oncol. 2022 Feb 1;8(2):242-250. doi: 10.1001/jamaoncol.2021.6268. PMID 34913959